CLINICAL TRIAL: NCT04317365
Title: Effect of Counseling Between Pregnant Women During Corona Infection
Brief Title: Counseling of Pregnant Women During Corona
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Respiratory infection
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients receiving remembering (Active Comparator)
  Interventions: Other: Women receiving extra remembering by healthcare
- patients not receiving extra remembering (No Intervention)

INTERVENTIONS:
Other: Women receiving extra remembering by healthcare — Women receiving extra remembering by healthcare in covid infection
  Arms: patients receiving remembering

SUMMARY:
Corona virus is known as covid 19 And is transmitted through droplet infection

DETAILED DESCRIPTION:
Symptoms of Corona include cough Fever and dyspnea

ELIGIBILITY:
Inclusion Criteria:

* pregnant women

Exclusion Criteria:

* non pregnant women

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 200 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
The number of pregnant women who know the exact symptoms of the disease | Within one month
  The number of pregnant women who have awareness about the disease

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Study Chair — Algezeera hospital
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt